CLINICAL TRIAL: NCT05139173
Title: User Centred Design and Pilot Testing of a Novel Shoulder Rehabilitation Program With Engagement Tracking
Brief Title: Novel Shoulder Rehabilitation Program (SPARS-REHAB)
Acronym: SPARS-REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARS-REHAB
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Pathology
Keywords: Rehabilitation; Artificial Intelligence; Wearable Electronic Devices; Adherence; Physiotherapy; Rotator Cuff Pathology

STUDY DESIGN:
Intervention Model Description: Device: Smart Physiotherapy Activity Recognition System (SPARS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Injured Worker Population (Experimental): Participants that have a confirmed rotator cuff pathology, and are undergoing physiotherapy at the Holland Centre for a work-related shoulder injury as part of the Working Condition Program.
  Interventions: Device: Smart Physiotherapy Activity Recognition System (SPARS)
- Active Comparator: OHIP (funded) Patient Population (Active Comparator): Participants that have a confirmed rotator cuff pathology, and are undergoing physiotherapy at the Holland Centre as part of the Shoulder Program.
  Interventions: Device: Smart Physiotherapy Activity Recognition System (SPARS)

INTERVENTIONS:
Device: Smart Physiotherapy Activity Recognition System (SPARS) — Wearable smart watch that records inertial data such as (accelerometer, gyroscope magnetometer) and the exercise is started on the tablet, while patients are performing physiotherapy exercises.

SUMMARY:
Physical therapy is essential for the successful rehabilitation of common shoulder injuries and following shoulder surgery. Patients may receive some training and supervision for shoulder physiotherapy through private pay or private insurance, but they are typically responsible for performing most of their physiotherapy independently at home. It is unknown how often patients perform their home exercises, if these exercises are done correctly without supervision, and how poor adherence might impact recovery.

The investigators have recently developed a Smart Physiotherapy Activity Recognition System (SPARS) for tracking home shoulder physiotherapy exercises using sensors in a commercial smart watch and artificial intelligence (AI). SPARS was successful in identifying shoulder exercises in healthy adults in the laboratory setting, and in patients undergoing physiotherapy for rotator cuff pathology. Further inquiry is required to establish the clinical effectiveness of this technology for tracking and improving patient engagement, and to investigate the potential individual impacts of its use.

DETAILED DESCRIPTION:
The Research Team will conduct in-person data collection on 30 patients, by recording patients' exercises during their supervised physiotherapy sessions each week using the SPARS smart watch. Each patient will wear the smart watch on their affected arm only when performing prescribed exercises, and the watch will start recording inertial sensor data once the patient puts the watch on and the exercise is started on the tablet. An app installed on the provided Android smart tablet allows the patient to view their assigned exercises, videos showing them how to perform those exercises, and the record of their tracked participation. A tablet app will also be available to the treating physiotherapist to allow them to view this same data. The purpose of the participation tracking is to promote better patient engagement in the home component of physiotherapy.

The injured worker population will be recruited from referrals made to the Sunnybrook Working Condition Program (WCP) at the Holland Centre for a work-related shoulder injury. Physical therapy of the patient population will be recruited from referrals by the Sunnybrook Shoulder and Upper Extremity Program funded by study grants. Data collection will be collected at each supervised physiotherapy session during the course of a patient's treatment. Follow-up outcomes such as surveys and shoulder testing will be done at 6 weeks, monthly at a maximum of 3 months (OHIP-patients) and 5 months (WSIB) patients, final treatment session (if different than maximum amount), and 1 year after.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females over the age of 18
2. Diagnosed with rotator cuff tendinosis, shoulder impingement syndrome, or degenerative or traumatic rotator cuff tear
3. Planned conservative (non-operative) management
4. Capacity to participate in home shoulder physiotherapy

Exclusion Criteria:

1. Upper extremity neurologic deficit
2. Symptomatic contralateral shoulder with limited mobility requiring treatment
3. Failed surgical management of rotator cuff pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Physiotherapy participation (Minutes weekly physiotherapy) | Up to 3-5 months
  Investigators will recruit up to 30 patients with rotator cuff pathology. Watch will begin recording inertial sensor data when it is put on by a patient during supervised and home physiotherapy exercises and the exercise is started on the tablet, and will stop recording when it is removed and the exercise is stopped on the tablet. Inertial data will be analyzed to generate quantitative measures of at-home physiotherapy participation in comparison to each patient's current physiotherapy prescription. Participation will be measured in minutes of weekly physiotherapy participation. Participation measurement will be compared to historical controls to detect statistically significant differences resulting from the use of apps by patients and their physiotherapists.

SECONDARY OUTCOMES:
Work status | Up to 1 year
  Clinical and return to work outcome data full-time, part-time, off-work, modified or regular duties.
Numeric Pain Rating Scale (NPRS) | Up to 1 year
  Scale range: 0 to 10 (whole number integers). Higher scores represent more pain.
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | Up to 1 year
  Self administered questionnaire to self rate upper extremity disability and symptoms. Comprises of a 30-item disability/symptom scale, and higher scores represent more symptoms/disability.
The American Shoulder and Elbow Society (ASES) Score | Up to 1 year
  Self administered questionnaire to self rate current shoulder pain and the ability to do 10 activities, and lower scores represent more inability to perform these activities.
Strength testing | Up to 12 weeks
  Rotator cuff strength testing using manual muscle testing as well as strength testing with a dynamometer.
Shoulder active range of motion | Up to 12 weeks
  Measured by a handheld goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Helen Razmjou, Principal Investigator — Sunnybrook Holland Orthopaedic & Arthritic Centre
Locations (1):
- Sunnybrook Holland Orthopaedic & Arthritic Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No